CLINICAL TRIAL: NCT00288314
Title: Working Memory Updating in Posttraumatic Stress Disorder (PTSD): Study of Neural Correlates Using fMRI
Brief Title: fMRI in Posttraumatic Stress Disorder (PTSD) During Working Memory Updating
Acronym: METRAPI
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: PHRR, CHRU TOURS
Other Study IDs: PHRR04-WEH/METRAPI
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Post-Traumatic Stress Disorders; Anxiety; Amnesia, Dissociative
Keywords: PTSD; MRI, Functional; Anxiety; Working Memory; Processing speed
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Amnesia | interventions — Magnetic Resonance Spectroscopy; Functional Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PTSD
  Interventions: Procedure: Magnetic Resonance Imaging, Functional
- CONTROLS
  Interventions: Procedure: Magnetic Resonance Imaging, Functional

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging, Functional — Structural and functional MRI

SUMMARY:
Neuropsychological studies investigating trauma-exposed and posttraumatic stress disorder (PTSD) subjects have generally underlined the significantly poorer performance of tasks that require attention, concentration, and verbal memory, and difficulty in regulating memories surrounding the traumatic event. A previous study (El Hage et al. Cognitive Neuropsychiatry, 2006) revealed that the trauma-exposed subjects scored higher on anxiety/depression scales, and lower on processing speed tests. Moreover, the study showed significant impairment in working memory partially mediated by speed processing, but not by anxiety or depression. These results suggest that processing speed makes a major contribution to trauma-related working memory decline, and needs to be investigated in further studies.The aim of the present study is to explore correlation between hippocampus volume, frontal dysfunction and cognitive slowing in trauma-exposed subjects, while examining brain activation during performance of working memory tasks using functional magnetic resonance.

DETAILED DESCRIPTION:
Working memory performance will be assessed using the "3-back test", and processing speed evaluated with "words comparison test". The study will be conducted on 2 years. The study should include 18 right-handed females victims of sexual abuse and suffering from PTSD, and 18 controls right-handed females without any history of abuse ad not suffering from PTSD. Brain activation will be measured during performance of working memory tasks (3-back test) and processing speed test using functional magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed women
* Victim of sexual abuse
* Suffering from PTSD

Exclusion Criteria:

* Epilepsy
* Claustrophobia
* MRI contre-indication
* Addictive disorders
* Sightless
* Detection of a brain injury at the MRI

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: PTSD related to sexual abuse vs controls, in right-handed females.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wissam EL HAGE, MD, PhD, Principal Investigator — UNIVERSITY HOSPITAL OF TOURS
Locations (1):
- University Hospital of Tours, Tours, Centre-Val de Loire, France

REFERENCES:
- [Background] El-Hage W, Gaillard P, Isingrini M, Belzung C. Trauma-related deficits in working memory. Cogn Neuropsychiatry. 2006 Jan;11(1):33-46. doi: 10.1080/13546800444000164. PMID 16537232